CLINICAL TRIAL: NCT05624866
Title: Dexmedetomidine Versus Triamcinolone Local Injection for Pain Alleviation in Patients With Carpal Tunnel Syndrome; A Randomized Clinical Trial.
Brief Title: Dexmedetomidine Versus Triamcinolone Treatment in Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17200681
Record Dates: First submitted 2022-10-31; First posted 2022-11-22 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-11

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Dexmedetomidine; Triamcinolone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Investigate if, and to what extent,carapl tunnel hydro-dissection using DEX or triamcinolone (TM) along with saline, under ultrasound guidance, can improve the clinical condition, change in nerve conduction parameters of patients with CTS and delay or avoid the surgical intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmeditomidine group (Active Comparator): injection of 1 microgram/kg dexmeditomidine + 10 cc saline injection nearby median nerve as hydro-dissection
  Interventions: Drug: Dexmedetomidine
- Triamcinolone group (Active Comparator): injection of 40 mg triamcinolone + 10 cc saline injection nearby median nerve as hydro-dissection
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Dexmedetomidine — injection of 1 microgram/kg dexmeditomidine + 10 cc saline injection nearby median nerve as hydro-dissection
  Arms: Dexmeditomidine group
Drug: Triamcinolone — injection of 40 mg triamcinolone + 10 cc saline injection nearby median nerve as hydro-dissection
  Arms: Triamcinolone group

SUMMARY:
Carpal tunnel syndrome (CTS) is a common mononeuropathy due to entrapment of the median nerve in the carpal tunnel. a lot of modalities are available for treatment of mild to moderate CTS.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a common mononeuropathy due to entrapment of the median nerve in the carpal tunnel. a lot of modaleties are available for treatment of mild to moderate CTS.

In case of failed conservative oral therapey, local hydro-dessction of the median nerve can be done with saline alone. local anethetics, steroids, hyalase,and ozone have been utilized to augment the symptoms reliefe.

Dexmeditomidine (DEX) has been studied as adjuvant for nerve block to aumnet the pain reliefe. Recently, it has been discovered that DEX can offer some antinflammatory effects when injected in the perineural area. Upon such discovery, the goal of this study has been built.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* complaining of carpal tunnel syndrome of 3 month duration or more
* diagnosed axonal neuropathy using electrodiagnosis , nerve conduction study

Exclusion Criteria:

* patient refusal
* infection at the site of intervention
* allergy to utilized drugs
* diabetic
* previous surgery in the site of injection
* previous injection in the targeted site within the last year

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
pain visual analoge scale visual analog scale of pain value of (0 cm) no pain , and value of (10 cm) worst pain | 6 months
  visual analog scale of pain value of (0 cm) no pain , and value of (10 cm) worst pain

SECONDARY OUTCOMES:
change of cross sectional area of the median nerve | 6 months
  change of cross sectional area of the median nerve mm2

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Universit Hospital, Asyut, Egypt